CLINICAL TRIAL: NCT03573375
Title: Cancer Patients' Reported Frequency and Barriers to Physical Activity
Brief Title: Barriers Affecting Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0993; NCI-2018-01526 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Cancer Patients and Physical Activity
Keywords: Questionnaires; Surveys
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer Patients in Supportive Care Clinic (SCC) (Experimental)
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete a series of questionnaires about exercise, symptoms, and physical abilities. These should take about 5 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this research study is learn about how often cancer patients engage in physical activity using the exercise behavior questionnaire.

This is an investigational study.

Up to 200 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
If participant agrees to take part in this study, participant will complete a series of questionnaires about exercise and participant's symptoms and physical abilities. These should take about 5 minutes to complete.

Additionally, demographic information (such as participant's age, race, sex, zip code, specifics about participant's cancer type and care) will be collected from participant's medical record.

Participant will complete the questionnaires 1 time, and participation in this study will be over after that.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 years of age or older.
2. Patient must be able to understand, read, write and speak English.
3. Patient must be able to sign an Informed Consent Form.

Exclusion Criteria:

1. Patients with physical limitations (visual, cognitive, motor impairment) causing inability to read, complete or sign the consent form and survey.
2. Wheelchair bound patients who spend all of their day in bed or wheelchair
3. Patients who the attending physician deems unable to participate due to acute physical distress.
4. Previously filled out (EBBS and Stanford) surveys in the Supportive Care Clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Cancer Patients Who Report Engaging in Physical Activity Using the Stanford Patient Education Research Center Exercise Behaviors Survey | 1 day
  Patients who report activity 1-3 hrs per week in any of the 6 questions or combination of any of these 6 questions are considered as engaging in physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org